CLINICAL TRIAL: NCT07019389
Title: Assessment of the Validity and Reliability of the Turkish Adaptation of the Child- and Parent-Rated Scales of Food Allergy Anxiety (SOFAA)
Brief Title: Validation of Turkish Versions Child- and Parent-Rated Scales of Food Allergy Anxiety
Status: Enrolling by invitation | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Hilal Gungor, Medical Doctor, Clinical Fellow in Pediatric Allergy and Immunology, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: b.30.2.ODM.0.20.08/111
Record Dates: First submitted 2025-06-04; First posted 2025-06-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Food Hypersensitivity; Allergy; Phobic Disorders; Caregiver Burden; Validation Study; Cross-Cultural Comparison; Parents; Anxiety; Pediatrics
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity; Phobic Disorders; Caregiver Burden; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Food Allergy: Children aged 8 to 18 years diagnosed with IgE-mediated food allergy, recruited from pediatric allergy clinics. Participants complete the Turkish-translated child version of the Scale of Food Allergy Anxiety (SOFAA-C).
  Interventions: Other: Turkish Version of the Scale of Food Allergy Anxiety (SOFAA)
- Parents of Children with Food Allergy: Parents or primary caregivers of the participating children complete the parent version of the Turkish-translated Scale of Food Allergy Anxiety (SOFAA-P)
  Interventions: Other: Turkish Version of the Scale of Food Allergy Anxiety (SOFAA)

INTERVENTIONS:
Other: Turkish Version of the Scale of Food Allergy Anxiety (SOFAA) — Participants will complete the Turkish-translated versions of the Scale of Food Allergy Anxiety (SOFAA). Children will complete the SOFAA-C; their parents will complete the SOFAA-P. The study aims to evaluate the reliability and validity of the translated scales through internal consistency, factor analysis, and test-retest reliability methods.

SUMMARY:
This study aims to evaluate the psychometric properties of the Turkish adaptation of the Scale of Food Allergy Anxiety (SOFAA), including both the child-report and parent-report versions. The SOFAA is a validated tool originally developed to assess the specific anxiety related to food allergies. The Turkish versions of the scales will undergo a comprehensive validation process, including assessments of internal consistency, test-retest reliability, and construct validity.

Participants will include children diagnosed with IgE-mediated food allergies and their primary caregivers. The study will investigate whether the translated scales maintain the original structure and effectively measure food allergy-related anxiety in the Turkish pediatric population. The findings are expected to contribute to clinical assessment practices and research on food allergy-related psychosocial impacts in Turkeyy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IgE-mediated food allergy
* At least one parent/caregiver willing to participate
* Fluent in Turkish

Exclusion Criteria:

* Major neurodevelopmental or psychiatric disorders that impair ability to complete scales

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 8-18 with food allergy and their parents, recruited from pediatric allergy outpatient clinics in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency of the Turkish Version of the SOFAA-C and SOFAA-P | Within 1 week of initial administration
  Internal consistency of the Turkish child- and parent-reported versions of the Scale of Food Allergy Anxiety (SOFAA) will be evaluated using Cronbach's alpha coefficient. A value of ≥ 0.70 will be considered acceptable.
Construct Validity of the Turkish Version of SOFAA | Within 1 week of initial administration
  Construct validity of the Turkish version of the SOFAA will be assessed using exploratory and/or confirmatory factor analysis based on responses from children and parents. Factor structure will be compared with the original version.
Test-Retest Reliability of the Turkish Version of SOFAA | Approximately 10-14 days after baseline assessment
  A subsample of participants will complete the SOFAA again after a 10-14 day interval. Test-retest reliability will be evaluated using intraclass correlation coefficient (ICC).

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Only aggregate results (e.g., internal consistency coefficients, summary statistics) will be shared. Individual participant data (IPD), even in de-identified form, will not be made publicly available. Access to data may be considered upon reasonable request and with appropriate ethical approvals.
Supporting Information: CSR
Time Frame: Aggregate data will be available beginning 6 months after study completion and for a period of up to 5 years thereafter.
Access Criteria: Researchers with a methodologically sound proposal may request access to the aggregated study data. Requests should be submitted to the principal investigator and will require appropriate ethical approval and a signed data-sharing agreement.

REFERENCES:
- [Background] Protudjer JLP. Scales of Food Allergy Anxiety (SOFAA): A Novel Tool to Assess Anxiety Among Children with Food Allergy and Their Caregivers. J Allergy Clin Immunol Pract. 2022 Jan;10(1):170-171. doi: 10.1016/j.jaip.2021.10.036. No abstract available. PMID 35000731
- [Background] Dahlsgaard KK, Wilkey LK, Stites SD, Lewis MO, Spergel JM. Development of the Child- and Parent-Rated Scales of Food Allergy Anxiety (SOFAA). J Allergy Clin Immunol Pract. 2022 Jan;10(1):161-169.e6. doi: 10.1016/j.jaip.2021.06.039. Epub 2021 Jul 12. PMID 34265450